CLINICAL TRIAL: NCT01640106
Title: Feasibility of Omega-3 Fatty Acid Supplementation for Children With Early Developmental Impairment in Language
Brief Title: Feasibility of Omega-3 Supplementation for Children With Language Impairments
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Recruitment very difficult; only preliminary data usable.
Sponsor: Shuvo Ghosh (Other)
Responsible Party: Sponsor-Investigator, Shuvo Ghosh, Assistant Professor of Pediatrics, McGill University Health Centre/Research Institute of the McGill University Health Centre
Organization: McGill University Health Centre/Research Institute of the McGill University Health Centre (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 09-164-PED
Record Dates: First submitted 2012-06-26; First posted 2012-07-13 (Estimated); Last update posted 2019-09-09 (Actual); Status verified 2019-09

CONDITIONS: Language Impairment
Keywords: Language; Fatty acids; Nutrition; Developmental delay
MeSH Terms: conditions — Language Disorders; Language; Learning Disabilities | interventions — Docosahexaenoic Acids

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Omega-3 (Experimental): Treatment arm, using the omega-3 product (fish oil/paste)
  Interventions: Dietary Supplement: Omega-3
- Control (Placebo Comparator): Placebo is a paste of non-omega-3 (plant based) oil with a taste/flavour identical to intervention paste
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Omega-3 — 800 mg Omega 3 daily (600 mg DHA/200 mg EPA)
  Other Names: Concordix chewable paste
  Arms: Omega-3
Dietary Supplement: Placebo — Placebo is a combination of dietary plant-based oils in a paste containing no Omega-3 (EPA or DHA)
  Arms: Control

SUMMARY:
The primary objective of this study is to obtain preliminary (pilot) data regarding the feasibility of using dietary omega-3 supplementation in children with significant delays in language skills; a related secondary objective is to compare adherence to a dosage schedule of two easy-to-take formulations. A tertiary objective of this study is to collect preliminary (pilot) data pre- and post-supplementation to identify potential improvement of skills in a specific area of language development.

DETAILED DESCRIPTION:
HYPOTHESIS Hypothesis 1: Children with early developmental impairment in language will successfully take daily omega-3 fatty acid supplementation for a well-defined period of time (3 months); Hypothesis 2: Children with early developmental impairment will better adhere to administration of a small quantity of slightly fishy-tasting oil than to a large quantity of sweet-tasting paste; Hypothesis 3: A 3 month period of daily omega-3 supplementation will produce some improvement in fast-mapping language skills (a dynamic vocabulary learning skill that has been shown to rapidly improve after exposure to beneficial intervention).

ELIGIBILITY:
Inclusion Criteria:

* children in the chronological age range of 24 to 42 months at the time of initial assessment
* diagnosis of expressive, receptive or mixed language impairment (LI) by a certified Speech-Language Pathologist (S-LP)
* ability to take daily omega-3 supplementation (with caregiver assistance)

Exclusion Criteria:

* children with any organic disease processes or genetic syndromes, or known developmental disorders such as autism that may present with language impairment
* children with hearing impairment
* children who take any non-standard dietary supplements (i.e., apart from multi-vitamins), particularly any omega-3 FA, prior to starting the study
* children whose parents do not have an adequate understanding of English or French

Ages: 24 Months to 42 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 8 (Actual)
Dates: Start 2012-06; Primary Completion 2014-03 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Change over 3 months in learning assessed by a fast-mapping task | Assessed at time of diagnosis and 3 months after intervention
  A simple "fast-mapping" task, which is a measure of language learning used widely in linguistics research, will be performed in the pre and post-intervention period. We will present a list of non-words selected with only early-developing sounds to ensure that they are within the repertoire of developmentally impaired children. Scores are calculated in terms of number of items successfully completed. An initial and final assessment of dynamic language learning will be done as an addendum to scores on standardized language tests that establish a language impairment diagnosis.

SECONDARY OUTCOMES:
Feasibility of fish oil vs. chewable Concordix paste | Given for 3 months as intervention
  In order to estimate the relative success of administering paste vs. oil in relation to omega-3 vs. placebo, a repeated measures ANOVA will be used to test for significant differences. The primary measure will be parental report as "easy" vs. "difficult" to administer, and the analysis will be run as Between group (paste vs. oil) by Treatment arm (omega-3 vs. placebo) by Adminstration success (easy vs. difficult).

CONTACTS AND LOCATIONS:
Overall Officials: Shuvo Ghosh, MD, Principal Investigator — MUHC Montreal Children's Hospital
Locations (1):
- McGill University/Montreal Children's Hospital, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: Undecided